CLINICAL TRIAL: NCT06636916
Title: Time at VO2max During High-Intensity Interval Training Manipulating Work and Rest
Brief Title: Time at VO2max During High-Intensity Interval Training
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maia (Other)
Responsible Party: Principal Investigator, Filipe Silvano Pinto Maia, Principal investigator, University of Maia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: _HIIT_FMJB
Record Dates: First submitted 2024-10-03; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: High Intensity Interval Exercise (HIIE)
Keywords: sports; hiit; athletic performance; vo2max

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- short intervals (Experimental): This group will perform the hiit by doing short intervals
  Interventions: Procedure: Short Intervals HIIT; Procedure: Long intervals HIIT
- long intervals (Experimental): This group will perform the hiit by doing long intervals
  Interventions: Procedure: Short Intervals HIIT; Procedure: Long intervals HIIT

INTERVENTIONS:
Procedure: Short Intervals HIIT — Participants will undergo different high-intensity interval training (HIIT) protocols, which involve repeated bouts of exercise at an intensity above 90% of VO2max, followed by recovery periods. The work and rest durations will vary across the protocols to assess the impact on the total time spent at or above 90% of VO2max.
Procedure: Long intervals HIIT — Participants will undergo different high-intensity interval training (HIIT) protocols, which involve repeated bouts of exercise at an intensity above 90% of VO2max, followed by recovery periods. The work and rest durations will vary across the protocols to assess the impact on the total time spent at or above 90% of VO2max.

SUMMARY:
The project titled "Time at VO2max During High-Intensity Interval Training Manipulating Work and Rest" aims to investigate how different high-intensity interval training (HIIT) protocols influence the time athletes spend at or above 90% of their VO2max. By adjusting the work-to-rest ratios in the HIIT formats, the study seeks to determine which configurations maximize the time spent in this high-intensity zone, contributing to more effective endurance training strategies. The findings could help optimize training protocols for athletes targeting improvements in aerobic capacity and performance.

ELIGIBILITY:
Inclusion Criteria:

* Middle and long distance track and field athletes

Exclusion Criteria:

* Injured athletes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
time above 90% vo2max | Duration of the HIIT (up to 20 minute)

IPD SHARING:
Plan to Share IPD: Undecided